CLINICAL TRIAL: NCT04514809
Title: Comparison of Milk Compositions of Tandem Breastfeeding Mothers With Milk Compositions of Single Infant Breastfeeding Mothers: Randomized Controlled Trial
Brief Title: Milk Compositions of Mothers Who Breastfeed as Tandem
Acronym: Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Nursan Cinar, Proffesor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Nursan CİNAR
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Tandem Breastfeeding
Keywords: Breastfeeding in pregnancy; tandem breastfeeding; human milk composition

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: The statistician was also blinded for the data analysis purpose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): It consists of 15 mothers who meet the inclusion criteria
  Interventions: Other: human milk analized
- Control Groups (Experimental): It consists of 15 mothers who meet the inclusion criteria
  Interventions: Other: human milk analized

INTERVENTIONS:
Other: human milk analized — After birth (24-72 hours) 15 ml, and end of the first month of birth 30 ml of milk from the mother will be milked in the appropriate way and put into the sterile milk collection container. The milk taken into the milk transport container will be delivered to the Nutrition Lab for analysis (moisture, protein, fat, lactose) by the researcher who arrives at the TUBITAK Mam Research Center as fresh within 3 hours

SUMMARY:
The impact of tandem breastfeeding on the health of mothers and babies is a matter of curiosity. It is stated in the literature that there are few studies that examine the results of tandem breastfeeding in terms of mother, newborn and other baby after birth, and that there are no negative consequences of breastfeeding in terms of mother, newborn and older baby at two different ages. Research shows that while it is possible for mothers to continue breastfeeding by counselling to them based on evidence-based information, most of them have ended breastfeeding. It is the responsibility of nurses to make this process more successful and seamless for both mothers and babies. In tandem breastfeeding, the nurse should advise the mother on her own feeding and breastfeeding, and should refer her to her physician if she considers it necessary. There is no clear and up - to-date source showing changes in mother's milk over time (24-72 hours-one month), production time (colostrum and mature milk), changes in milk composition in tandem breastfeeding in the current literature, and this study is original with this aspect.

DETAILED DESCRIPTION:
Background: Considering the health benefits both for the infant and the mother, American Academy of Pediatrics (AAP) and World Health Organization (WHO) recommend only mother's milk in the first six months of life and then continuing breastfeeding for at least two years with complementary feeding (Eidelman, 2012; Topal et al., 2011). A review of the breastfeeding status of babies in Turkey reveals that breastfeeding is common, but it is not at a satisfactory level in terms of the length of time babies are given mother's milk only or in the total length of breastfeeding. One of the most important reasons is early start of complementary food or early weaning (TNSA2018). In 5.7 to 29.2% of the cases where breastfeeding was terminated early, the mother became pregnant again during the lactation period. Both mothers and healthcare professionals are confused as to whether breastfeeding should continue in pregnancy. Moreover, the field literature does not offer any information about any changes in the milk composition of a mother breastfeeding two babies of different ages at the same time (tandem breastfeeding). It is also known that some mothers who get pregnant during lactation period or with an interval of less than two years do not wean the first-born and continue breastfeeding both babies at the same time (Bøhler & Ingstad, 1996; Moscone & Moore, 1993; O'Rourke & Spatz, 2019). In light of this information, this study project is aimed to explore any differences in the composition (fat, protein, lactose, water, and casein) and density of milk during pregnancy or tandem breastfeeding.

Method: The universe of the study is planned to consist of all multigravid women admitted to the Obstetrics and Gynecology Clinic of the Sakarya University Education and Research Hospital, Turkey, breastfeeding postpartum in tandem and not breastfeeding during pregnancy. The sample of the study, including 15 control and 15 experimental groups, 30 mothers to be selected according to the inclusion criteria. groups will be determined by simple random sampling method. In order to assign the mothers who meet the selection criteria into the experimental group or the control group, the randomization method with a computer program (http://www1.assumption.edu/users/ avadum/applets/RandAssin/Groupgen.html) was used. Data collection is planned to take place in two stages for control and experimental groups. The first stages correspond to 24 to 72 hours postpartum. This is to be accomplished through house calls upon appointment with the mothers. During the house call, 15 ml milk is obtained from the mother with suitable methods (Appendix…) and preserved in a sterilized milk collection container. At the end of birth, 15 ml colostrum will be taken from the mother, instead of 30 ml, so that the babies in both groups benefit more from colostrum. Then, it is analyzed within the next 3 hours in terms of its composition (moisture, protein, oil, lactose) and to the Tubitak Mam Research Center to the Nutrition Lab for analysis.Results are recorded in the "Breastfeeding Follow-up Form." The final stages (after the 1st month postpartum), during the house call, 30 ml milk is obtained from the mother with suitable methods (Appendix…) and preserved in a sterilized milk collection container, other steps will be repeated in the same order. The results of the analysis will be compared with the breast milk compositions in the control group. The results of this study are expected to clarify the attitudes of healthcare professionals about tandem breastfeeding and to draw attention to this issue, thereby providing guidance and encouragement for further studies on the subject..

ELIGIBILITY:
Inclusion Criteria:

Being mature newborn (<37 GW) Being a mother who in third trimester The mother's lack of a health problem from a metabolic and endocrine perspective related to nutrition Absence of diagnosed psychiatric story of the mother Mother's openness to communication and cooperation Mother's volunteering to participate in the study Mother being literate Having multigravida of the mother Mother's age above 18 years Being a mother non-vegetarian Being a mother non-smoker Absence of breast trauma in mother (mastitis, abscess etc.) Mother's milk analysis at least a week before without taking any medication Having body mass index at normal values (18.5 to 24.9) pre-pregnancy (WHO, 2015).

Exclusion Criteria:

Having a condition that obstacle for breastfeeding (craniofacial abnormality such as cleft palate, cleft lip, paralysis of facial muscles)

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the protein level of breast milk in study and control groups | 24 to 72 hours postpartum and of the 1st month postpartum
  The measurement values will be recorded on the "mother milk follow form" which was created by the researchers.
Evaluation of breast milk fat level in study and control group | of the 1st month postpartum
  The measurement values will be recorded on the "mother milk follow form" which was created by the researchers
Evaluation of lactose level of breast milk in study and control group | of the 1st month postpartum
  The measurement values will be recorded on the "mother milk follow form" which was created by the researchers.
Evaluation of moisture level of breast milk in study and control group | of the 1st month postpartum
  The measurement values will be recorded on the "mother milk follow form" which was created by the researchers.

SECONDARY OUTCOMES:
Feeding follow-up of mothers | 24 to 72 hours postpartum and the 1st month postpartum
  This form is the form in which the participants recorded all the nutrients they had consumed in the last three days as six meals, with three main and three intermediates. Information will be provided to the participants by the researcher (O.K.S.) about how to record the amounts of all the food and drink they consumed in the last three days with standard sizes such as units, numbers, grams, water or tea cups, cups, etc. Forms will be distributed in order to record all the nutrients they consume in the same day regularly as meals and collected back on home visit days. With this form, the daily consumption amounts of energy, vitamins, minerals, protein, fat, carbohydrates, fiber and beverages will be analyzed in the nutrition information system (Bebis 8.0) software package program.

CONTACTS AND LOCATIONS:
Overall Officials: Nursan Cinar, PhD, Study Director — Sakarya University; özge suzan, Msc, Principal Investigator — Sakarya University; serhan cevrioglu, PhD, Principal Investigator — Sakarya University

IPD SHARING:
Plan to Share IPD: No